CLINICAL TRIAL: NCT06792734
Title: Phase 1A/1B Trial of BTM-3566 in Relapsed/Refractory Mature B Cell Lymphomas
Brief Title: Phase 1 Trial of BTM-3566 in Relapsed/Refractory Mature B Cell Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bantam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTM-3566-001
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BTM-3566 Treatment (Experimental): BTM-3566 Oral Solution
  Interventions: Drug: BTM-3566

INTERVENTIONS:
Drug: BTM-3566 — Oral Solution
  Other Names: BTM-3566 Oral Solution

SUMMARY:
The goal of this clinical trial is to learn if BMT-3566 can safety be given to adult patients with relapsed or refractory mature b cell lymphomas. It will also learn how well BTM-3566 works to treat relapsed or refractory mature b cell lymphomas. The main questions it aims to answer are:

What are the side effects of BTM-3566 at different doses? What are the levels of BTM-3566 in the blood at different timepoints around dosing? What is the clinical benefit of BTM-3566 in treating cancer (i.e. how well does it slow or stop disease progression)?

Participants will:

Take BTM-3566 in 14-day periods with 7 days of dosing followed by 7 days of no dosing Visit the clinic regularly for checkups and tests Keep a diary of their dosing and weight

DETAILED DESCRIPTION:
This is an open label, phase 1 dose escalation trial of BTM-3566 in relapsed/refractory mature b cell lymphomas. Dose escalation will utilize traditional 3+3 methodology to determine the maximum tolerated dose of BTM-3566. Treatment will be given as two-week cycles, with BTM-3566 taken daily during the first week of the cycle, and the second week 'off therapy'. DLT window will be the first two cycles of therapy (days 1 to 28). All enrolled patients will undergo a baseline FDG-PET/CT scan within 3 weeks prior to starting therapy. FDG-PET/CT will be repeated at the start of Cycles 3 and 5 or more frequently as clinically indicated. Beginning at Cycle 5, imaging will be repeated every 3 months (or as clinically indicated) for up to 12 months, and every 6 months thereafter, until disease progression or start of subsequent anti-cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* must be age ≥18 years
* must have a diagnosis of relapsed or refractory mature B cell lymphoma
* must have measurable disease per response evaluation criteria in lymphoma (Lugano classification)
* must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* must have a predicted life expectancy of ≥3 months
* must agree to use adequate birth control throughout their participation and for 90 days following the last dose of BTM-3566

Exclusion Criteria:

* has primary CNS lymphoma
* has ongoing toxicities from prior anti-cancer treatment > Grade 1
* has symptomatic or uncontrolled neurologic disease (brain metastases, leptomeningeal disease, or spinal cord compression) not definitively treated with surgery or radiation
* has received any anti-cancer therapy (including radiation of curative intent) <28 days prior to administration of BTM-3566
* has current second malignancy at other sites (exceptions: non-melanomatous skin cancer, adequately treated in situ carcinoma, or indolent prostate cancer under observation).
* is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Event and dose-limiting toxicity event rates | 24 months
  The rate of adverse events and dose-limiting toxicity of therapy with BTM-3566

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Bashir, MBBS, Study Director — Bantam Pharmaceuticals
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No